CLINICAL TRIAL: NCT03654755
Title: A Phase 2, Multicenter, Open-Label Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of ASN002 in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Study to Evaluate Long-Term Safety of ASN002 in Subjects With Moderate to Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Phase 2 study results
Sponsor: Asana BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASN002AD-201-EXT
Record Dates: First submitted 2018-08-16; First posted 2018-08-31 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Atopic Dermatitis
Keywords: eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — gusacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ASN002 40 mg (Experimental): ASN002 40 mg
  Interventions: Drug: ASN002
- ASN002 60 mg (Experimental): ASN002 60 mg
  Interventions: Drug: ASN002
- ASN002 80 mg (Experimental): ASN002 80 mg
  Interventions: Drug: ASN002

INTERVENTIONS:
Drug: ASN002 — Daily dose of ASN002 for up to 110 weeks

SUMMARY:
This is a randomized open label study to evaluate the long term safety of ASN002 in subjects with moderate to severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
This is a randomized open label study where subjects with moderate to severe atopic dermatitis will roll over from the Phase 1 ASN002AD-101 (NCT03139981) and ASN002AD-201 (NCT03531957) Ph2b study and be randomized to receive ASN002 at 40mg, 60mg, or 80mg once daily for up to 24 months. This study will also characterize the pharmacokinetics of ASN002 through blood sampling from subjects who consent.

ELIGIBILITY:
Inclusion Criteria

* Subject with a history of moderate to severe atopic dermatitis who participated in the preceding ASN002AD-201 and ASN002AD-101 study
* Subject must be a candidate for prolonged open label ASN002/gusacitinib treatment according to the investigator's judgment.
* Subject has been using an emollient daily for at least 1 week prior to Day 1 and agrees to continue using that same emollient daily throughout the study.
* Men and women participating in the study must use medically acceptable birth control or total abstinence from sexual intercourse
* Subject is willing to participate and is capable of giving informed consent. Note: Consent must be obtained prior to any study-related procedures.
* Subjects must be willing to comply with all study procedures and must be available for the duration of the study.
* Subject has a body mass index (BMI) ≤ 38 kg/m2.

Exclusion Criteria

* Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
* Subject has clinically infected atopic dermatitis.
* A serious uncontrolled condition including hypertension, history of tuberculosis, hepatitis B or C infection, immune deficiency, heart disease, heart conduction disorder, diverticulitis, diabetes, reflux disease requiring protocol pump inhibitor therapy, malabsorption syndrome, or cancer
* Subject has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments.
* Subject has a history of eczema herpeticum within 12 months, and/or a history of 2 or more episodes of eczema herpeticum in the past.
* Willing to comply with discontinuation of certain treatments for AD, as directed by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Zammit, Ph.D., Study Director — Asana BioSciences
Locations (38):
- United States (31):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Total Skin and Dermatology Center, PC., Birmingham, Alabama
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - L.A. Universal Research Center, Inc., Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Revival Research, Doral, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Leavitt Medical Associates of Florida, Ormond Beach, Florida
  - Dermatology Consulting Services, Tampa, Florida
  - Forward Clinical Trials, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Dermatology Center of Indiana, PC, Plainfield, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Central Kentucky Research Associates, LLC, Lexington, Kentucky
  - Dermatology Specialists Research, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - ActivMed Practices and Research, Inc., Portsmouth, New Hampshire
  - Corning Center for Clinical Research, Corning, New York
  - Mt. Sinai Hospital, New York, New York
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Dermatologists of Greater Colombus, Bexley, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, Tulsa, Oklahoma
  - DermDox Centers for Dermatology, Hazleton, Pennsylvania
  - Synexus, Greer, South Carolina
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Innovate Research, LLC, Fort Worth, Texas
  - The Center for Skin Research, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Canada (7):
  - Institute of Skin Advancement Medical, Surgical, Costmetic & Laser Dermatology, Calgary
  - Innovaderm Research, Inc., Montreal
  - Ontario Inc., Ottawa
  - York Regional Dermatology, Richmond Hill
  - NewLab Clinical Research, Inc., St. John's
  - AvantDerm, Toronto
  - SkinWISE Dermatology, Winnipeg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from ASN002AD-101 and ASN002AD-201 were eligible to enter the OLE study if they (1) had participated in ASN002AD-101 study OR (2) had participated in ASN002AD 201 study, had completed at least the first 4 weeks without the use of prohibited treatments for AD, and had completed the study visits up to Week 12. Participants who had received the placebo in the other preceding studies were allowed to be enrolled in the OLE study except those who were responders at Week 12 based on EASI75
Pre-assignment Details: Those participants that received placebo in ASN002AD-201 or were enrolled in ASN002-101 were allocated as starting treatment, and those that received ASN002 in ASN002AD-201 trial are allocated as continuing treatment.
Period: Overall Study
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg
Started | 45 | 41 | 76
New Start of Treatment | 9 | 12 | 15
Continued Treatment (Continued treatment from parent study) | 36 (Includes 11 participants that started at 40 mg and received a dose escalation during the study) | 29 (Includes 6 participants that started at 60 mg and received a dose escalation to 80 mg during the study) | 61
Completed | 0 | 0 | 0
Not Completed | 45 | 41 | 76
Not completed — Early Termination of study due to COVID-19 | 42 | 33 | 56
Not completed — Withdrawal by Subject | 2 | 4 | 8
Not completed — Lost to Follow-up | 1 | 3 | 7
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg | Total
Number analyzed (Participants) | 45 | 41 | 76 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 35 | 69 | 143
  >=65 years | 6 | 6 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (18.34) | 42.3 (17.15) | 42.9 (15.9) | 42.4 (16.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 36 | 84
  Male | 19 | 19 | 40 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 5 | 2 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 8 | 7 | 11 | 26
  White | 32 | 31 | 57 | 120
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Eczema Area Severity Index (EASI) Score
Description: The Eczema Area and Severity Index (EASI) is a composite score ranging from 0 to 72, the higher the value the worse the disease, that takes into account the degree of erythema, induration/infiltration (papules), excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the percentage of BSA involved for each body region and for the proportion of the body region to the whole body.
  Due to early termination of the study, all efficacy analyses were descriptive in nature
Time Frame: 3 Months
Population: The number of participants analyzed includes those that had a 3 months time point assessed before early termination of the study. Therefore, the numbers analyzed are not the same as those that started or completed the study.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg
Number analyzed (Participants) | 22 | 18 | 42
Change in score on a scale | -22.88 (12.914) | -18.07 (7.687) | -17.38 (13.561)

2. Secondary Outcome: Number of Participants Achieving an Investigator Global Assessment (IGA) Scale of Clear (0) or Almost Clear (1)
Description: The IGA is a global assessment of the current state of the disease. It is a 5-point (0-4) morphological assessment of overall disease severity. The IGA is selected using descriptors that best describe the overall appearance of the lesions at any given point. Signs like inflammation, redness, oozing, and crusting are evaluated. The 0 is the least severe and 4 is the most severe.
  Due to early termination of the study, all efficacy analyses were descriptive in nature.
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg
Number analyzed (Participants) | 22 | 18 | 43
Participants | 8 | 8 | 9

3. Secondary Outcome: Change From Baseline in 5-D Pruritus (Itch) Scale
Description: The 5-D Pruritus Scale is a validated questionnaire used in clinical trials to assess the degree, duration, direction, disability, and distribution of the itch to rate the their symptoms over the preceding 2-week period. Each symptoms is scored on a scale of 1 to 5, with 5 being the most affected. The total score of 5-D pruritus is a sum of the 5 scores to provide a total score range from 5 (best) to 25 (worst).
  Due to early termination of the study, all efficacy analyses were descriptive in nature
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg
Number analyzed (Participants) | 22 | 18 | 43
change in score on a scale | -7.7 (4.21) | -7.1 (4.93) | -6.9 (4.97)

4. Secondary Outcome: Change From Baseline in Pruritus (Itch) Numeric Rating Scale (NRS)
Description: Intensity of itch will be measured using an NRS to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable" Due to early termination of the study, all efficacy analyses were descriptive in nature
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg
Number analyzed (Participants) | 19 | 18 | 40
change in score on a scale | -3.4 (2.99) | -3.3 (2.93) | -3.2 (3.16)

5. Secondary Outcome: Change From Baseline in Patient-Oriented Eczema Measure (POEM)
Description: POEM developed by Charman et al. is a self-assessment of disease severity by the participant. The POEM includes 7 questions to evaluate the number of days the signs and symptoms of eczema over the last week. The answer to each question is categorized by the frequency of the sign or symptom from no days to 7 days. Each question is scored from 0 to 4 and the sum of the questions if the POEM score. The score ranges from 0 to 28 with 0 being the least frequency and 28 showing that all the signs and symptoms occur every day. Therefore, the higher the score, the more severe the eczema. Due to early termination of the study, all efficacy analyses were descriptive in nature
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg
Number analyzed (Participants) | 22 | 18 | 42
change in score on a scale | -11.0 (7.04) | -11.5 (8.73) | -8.7 (8.08)

ADVERSE EVENTS:
Time Frame: Participants were to receive ASN002 once daily for up to 24 months. However, the study was early terminated approximately 12 months after initiation. The mean study treatment exposure ranged between 111.5 and 145.7 days, and the median ranged between 87.5 and 116.0 days
Groups:
- ASN002 40 mg: ASN002 40 mg
  Daily dose of ASN002
- ASN002 60 mg: ASN002 60 mg
  Daily dose of ASN002
- ASN002 80 mg: ASN002 80 mg
  Daily dose of ASN002
Arm/Group | ASN002 40 mg | ASN002 60 mg | ASN002 80 mg
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/41 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/41 | 1/76
Other Adverse Events (participants affected / at risk) | 2/45 | 3/41 | 6/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ASN002 40 mg (N=45) | ASN002 60 mg (N=41) | ASN002 80 mg (N=76)
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ASN002 40 mg (N=45) | ASN002 60 mg (N=41) | ASN002 80 mg (N=76)
Nasopharyngitis (Infections and infestations) | 1 | 3 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT03654755/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT03654755/SAP_001.pdf